CLINICAL TRIAL: NCT04873375
Title: Cemiplimab Treatment in Patients with Locally Advanced and Metastatic Secondary Angiosarcomas
Brief Title: Cemiplimab for Secondary Angiosarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Genzyme Europe B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-005465-13
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-06

CONDITIONS: Secondary Angiosarcoma; Locally Advanced Sarcoma; Metastasis
Keywords: Secondary Angiosarcoma; Cemiplimab; immunotherapy; Angiosarcoma; Sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Hemangiosarcoma; Sarcoma | interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: All patients included in this interventional single arm study will be treated with cemiplimab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cemiplimab (Experimental): After inclusion, all patients will be treated with Cemiplimab 350mg intravenously every three weeks
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — After inclusion patients will be treated with Cemiplimab 350mg intravenously every three weeks
  Other Names: LIBTAYO

SUMMARY:
Secondary angiosarcomas are aggressive mesenchymal tumors with a poor prognosis and limited therapeutic options. Recent studies conducted in patients with cutaneous squamous-cell carcinoma provide evidence that cemiplimab has the potential to be an effective treatment also for patients with secondary angiosarcomas.

The purpose of this study is to evaluate the overall response rate after 24 weeks of cemiplimab treatment in patients with locally advanced or metastatic secondary angiosarcomas.

The investigators hypothesis is that cemiplimab could be an effective treatment for patients diagnosed with locally advanced and metastatic secondary angiosarcomas.

DETAILED DESCRIPTION:
Study design: A prospective, interventional, non-randomized, multicenter, phase II clinical trial.

Hypothesis:

Cemiplimab is registered for the use in patients with cutaneous squamous-cell carcinoma. In these patient groups cemiplimab showed impressive results. There are numerous similarities between cutaneous squamous-cell carcinoma and secondary angiosarcomas. Based on these similarities, including a complex genetic background, PD-L1 expression and MYC expression, the investigators hypothesize that cemiplimab might be an effective treatment for locally advanced and metastatic secondary angiosarcomas.

Primary Objective:

To evaluate the overall response rate (ORR) after 24 weeks of cemiplimab in secondary angiosarcomas, according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 or daylight photography as per WHO Offset Publication No. 48.

Secondary Objectives:

Secondary objectives include the establishment of the best ORR, median time to response, duration of response and progression free survival. The secondary objectives also comprise safety and toxicity quantification and to investigate the relation between response to cemiplimab and various tumor characteristics.

Study Population:

Patients eligible for inclusion are at least 18 years of age, with adequate organ function, who have a histologically confirmed diagnosis of progressive unresectable locally advanced or metastatic secondary angiosarcoma. Patients eligible are patients in the first line of treatment if they are unfit for chemotherapy and patients in advanced lines of systemic treatment. Major exclusion criteria include significant ongoing autoimmune disease that requires immunosuppressive treatment, prior treatment with immune checkpoint inhibitors, active uncontrolled infections or recent pneumonitis. All patients will provide Informed Consent prior to inclusion in the study and during the course of the trial, al relevant data will be stored in electronic Case Report Forms (eCRF).

Treatment Schedule:

After study inclusion, patients will be treated with Cemiplimab 350mg intravenously every three weeks. Patients will receive treatment until disease progression or discontinuation due to unacceptable toxic effects, withdrawal of consent or other reasons. The maximum treatment period will be two years, as is standard of care for patients treated with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient aged ≥ 18 years.
2. Signed written informed consent.
3. Histologically confirmed diagnosis of progressive unresectable locally advanced or metastatic secondary angiosarcoma.
4. Patients in the first line of systemic treatment unfit for chemotherapy and patients in advanced lines of systemic treatment.
5. Measurable disease per RECIST 1.1 or per physical examination / daylight photography (WHO Offset Publication No. 48) as determined by the investigator.
6. Tumour tissue material available (archival or recent tumour biopsy).
7. WHO ECOG 0-2.
8. Hepatic function:

   1. Total bilirubin ≤ 1.5 x ULN (if liver metastases: ≤ 3 x ULN).
   2. Transaminases ≤ 3 x ULN (if liver metastases: ≤ 5 x ULN).
   3. Patients with Gilbert's Disease and total bilirubin up to 3x ULN may be eligible after communication with and approval from the medical monitor
   4. Alkaline phosphatase ≤ 2.5 x ULN (if liver OR bone metastases ≤5 x ULN).
9. Renal function: serum creatinine ≤ 2 x ULN or estimated CrCl > 30 mL/min.
10. Creatine phosphokinase (CPK) (also known as CK [creatine kinase]) elevation ≤ grade 2
11. Bone marrow function:

    1. Hemoglobulin ≥ 9.0 g/dL.
    2. ANC ≥ 1.5 x 109/L.
    3. Platelet count ≥ 75 x 109/L.
12. Expected life expectancy of at least 3 months as judged by the investigator.

Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for irAEs. The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 Diabetes mellitus, residual hypothyroidism that required only hormone therapy, or psoriasis that does not require systematic treatment.
2. Prior treatment with immune checkpoint inhibitors.
3. Continuous immunosuppressive corticosteroid treatment (doses > 10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of cemiplimab. Note: patients who require a brief course of steroids (e.g. as prophylaxis for imaging studies) are not excluded.
4. Active uncontrolled infection requiring therapy, including infection with HIV, active infection with HBV or HCV.
5. History of pneumonitis within the last 5 years.
6. Untreated brain metastasis(es) that may be considered active.

   a. Note in clarification: Patients with previously treated brain metastases may participate provided that the lesion(s) is (are) stable (without evidence of progression for at least 6 weeks on imaging obtained in the screening period), and there is no evidence of new or enlarging brain metastases, and the patients do not require any immunosuppressive doses of systemic corticosteroids for management of brain metastasis(es) within 28 days of the first dose of cemiplimab.
7. Patients with allergy or hypersensitivity to cemiplimab or to any of the excipients must be excluded. Specifically, because of the presence of trace components in cemiplimab, patients with allergy or hypersensitivity to doxycycline or tetracycline are excluded.
8. History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments
9. Patients with a history of solid organ transplant (patients with prior corneal transplants may be allowed to enroll after discussion with and approval from the medical monitor).
10. Any anticancer treatment other than radiation therapy (chemotherapy, targeted systemic therapy, imiquimod, photodynamic therapy), investigational or standard of care, within 30 days of the initial administration of cemiplimab or planned to occur during the study period
11. Receipt of live vaccines (including attenuated) within 30 days of first study treatment
12. Prior use of PI3K-D inhibitors
13. Women of childbearing potential (WOCBP)*, or sexually active men, who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment prior to the start of the first treatment, during the study, and for at least 6 months after the last dose.
14. Breastfeeding
15. Positive serum pregnancy test (a false positive pregnancy test, if demonstrated by serial measurements and negative ultrasound, will not be exclusionary, upon communication with and approval from the medical monitor)
16. Any other condition that might interfere with experimental treatment and the study procedures as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) after 24 weeks of cemiplimab | From the date of study inclusion until 24 weeks after inclusion. Interim analysis after 13 patients
  To evaluate the overall response rate (ORR) after 24 weeks of cemiplimab in secondary angiosarcomas, according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 or daylight photography as per WHO Offset Publication No. 48.

SECONDARY OUTCOMES:
Best Overall Response Rate | From the date of study inclusion to the end of the treatment period. Assessed up to 2 years after inclusion
  To establish the best ORR of patients with secondary angiosarcomas receiving cemiplimab
Time to response and duration of response | From the date of study inclusion to the date of response or progression. Assessed up to 2 years after inclusion
  To establish the median time to response (TTR) and duration of response (DOR) in patients with secondary angiosarcomas receiving cemiplimab.
Progression free survival (PFS) | Counting from the date of study inclusion to the date of progressive disease or death. Assessed up to 2 years after inclusion.
  To assess the median progression-free survival (PFS) of patients with secondary angiosarcomas receiving cemiplimab
Overall survival (OS) | From the date of study inclusion to the date of death. If study medication is discontinued for any reason, survival follow-up takes place every 12 weeks, also assessed up to 2 years
  To establish the overall survival (OS) of patients with secondary angiosarcomas receiving cemiplimab
Relation between tumor characteristics and response to treatment | 2-3 years
  To investigate possible relations between response to cemiplimab and tumor characteristics (i.e. PD-L1 expression, tumour infiltrating lymphocytes, MYC status and tumour mutational burden)
Differences between UV associated and radiation induced secondary angiosarcomas | 2-3 years
  To assess differences in response to cemiplimab between UV associated and radiation induced secondary angiosarcomas
Effect on tumor tissue | At specific timepoints tumor biopsies and liquid biopsies will be obtained. Tumor biopsies will be obtained at baseline, after 12 weeks and (voluntary) at end of treatment
  To assess effects of cemiplimab on tumor tissue by comparing pre- and post-treatment biopsies
Adverse events and toxicity | From the date of inclusion until the end of the study (by progression or at the end of the treatment period, up to 2 years
  To quantify toxicity during cemiplimab treatment

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes